CLINICAL TRIAL: NCT00370058
Title: Modulation of Homocysteine-Plasma Levels by ECT - Association With Clinical Response. A Pilot Study in Patients With Major Depression
Brief Title: Study on the Influence of Electroconvulsive Therapy (ECT) on Homocysteine Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECT and Homocysteine; Homocystein; ECT
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Depressive Disorder, Major
Keywords: ect; depression; homocysteine; mthfr genotype
MeSH Terms: conditions — Depressive Disorder, Major; Epilepsy, Rolandic; Depression

INTERVENTIONS:
Procedure: ECT treatment

SUMMARY:
Elevated homocysteine levels are associated with depression and cognitive impairment. When depression ameliorates due to treatment, homocysteine serum levels often normalize. Aim of the present study is to investigate, whether repeated ECT treatment leads to changes in homocysteine levels and if these changes are associated with the occurrence of cognitive impairment after ECS.

10 patients suffering from therapy-resistant depression shall be enrolled. Patients are treated with repeated ECT (three times the week). Before, directly after and one day after ECT treatment, blood samples are drawn and patients receive cognitive testing. Depressive symptomatology is checked with different rating scales.

DETAILED DESCRIPTION:
BACKGROUND:

Elevated homocysteine levels have been found in depressive disorders. The modulating effects of homocysteine on glutamatergic neurotransmission have been discussed to be an underlying cause of depression and can also lead to cognitive impairment and may facilitate seizures. Electroconvulsive therapy is the most effective treatment for depression, but often leads to cognitive impairments.

HYPOTHESIS:

Homocysteine levels normalize during rECT. This normalization is associated with the clinical improvement of depression. Short term changes in homocysteine levels (i.e. increase directly after ECT) may explain the cognitive impairments of the patients.

METHOD:

10 patients with therapy-resistant depressive disorder are to be enrolled into the trial. Patients are treated with rECT, two to three times a week. Blood withdrawal and psychometric analysis will be performed before, directly after and one day after ECT treatment 1,4,7,10,(13). Necessity of further treatment will be checked after the first 6 ECTs.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women aged 18 years or above
* Diagnosis of major depressive disorder (according to DSM IV)
* Secured therapy resistance (at least two trials with antidepressive medication of different classes for more then 4 weeks in adequate dosage)
* Written, informed consent

Key Exclusion Criteria:

* Major neurological or other diseases
* Current medication with antiepileptic drugs
* History of major head trauma
* Any medical condition not allowing anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Homocysteine serum levels

SECONDARY OUTCOMES:
Cognitive functioning (e.g. concentration, memory tasks, etc.)
Depressive symptomatology
Measures of Seizure quality (duration, threshold, postictal suppression index, ...)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bleich, M.D., Principal Investigator — University Erlangen-Nuremberg; Wolfgang Sperling, M.D., Study Director — University of Erlangen-Nürnberg
Locations (1):
- Department of Psychiatry and Psychotherapy, University Erlangen-Nuremberg, Erlangen, Germany